CLINICAL TRIAL: NCT02675972
Title: Association of 24-hour Blood Pressure Variability With Early Outcomes in Patients With Acute Non Cardiogenic Ischemic Stroke
Brief Title: Which Parameters of Short-term Blood Pressure Variability Best Predict Early Outcomes in Acute Ischemic Stroke
Acronym: BPV
Status: Completed | Type: Observational
Sponsor: Dongguan People's Hospital (Other Government)
Responsible Party: Principal Investigator, Zhu Shi, deputy director of neurology department, Dongguan People's Hospital
Other Study IDs: DongguanPeoplesH
Record Dates: First submitted 2016-01-27; First posted 2016-02-05 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Stroke
Keywords: stroke, blood pressure, prognosis
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — fasting glucose, creatine, BNP, CRP,BUN,cholesterol, LDL,HDL
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patient with poor outcome: modified Rankin scale≥3
- patients with favorable outcome: modified Rankin scale<3

SUMMARY:
Previous studies on the association between blood pressure variation (BPV) in acute ischemic stroke and functional outcomes yield conflicting result. The obscured definition and measurement of BPV engenders considerable confounding factors, making it difficult to interpret. We aim to investigate the predictive role of 24-hour BPV on early outcomes in acute non-cardiogenic ischemic stroke.

DETAILED DESCRIPTION:
This is a perspective registered cohort study. Patients with acute non-cardiogenic ischemic stroke are included into the study. During the first 24 hours after admission, the 24 hours blood pressure monitoring is to be taken and used to calculate various parameters of hour-to-hour blood pressure variability, including standard deviation(SD), coefficient of variation (CV), variation independent of mean(VIM) and average real variability (ARV) of systolic blood pressure (SBP) and diastolic blood pressure (DBP). The demographic and clinical data are also recorded. This is an observational sturdy, thus the caring physician make clinical decisions according to individual patient's condition. The endpoints are defined as early neurological deterioration, functional outcome(modified Rankin scale<3 as good outcome) at discharge and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* acute ischemic stroke

Exclusion Criteria:

* cardiogenic cerebral embolisms due to atrial fibrillation, pronounced heart valve diseases or valve replacement operation;
* isolated sensory symptoms, isolated visual changes, isolated dizziness, or vertigo, without explicit MRI-DWI evidence for acute cerebral infarcts;
* coexisting severe systematic diseases on admission such as acute coronary syndrome, malignant tumor, plasma dialysis therapy for renal failure, cirrhosis, rheumatic disease which would influence patients' independent functions .

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: acute ischemic stroke patients with 72 hour after onset
Sampling Method: Non-Probability Sample
Enrollment: 260 (Actual)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
early neurological deterioration | 7 days after admission
  NIHSS increase by 4 points or continuous consciousness deterioration

SECONDARY OUTCOMES:
good functional outcome at 14 days | up to 14 days in-hospital
  good functional outcomes as mRS≤2; poor outcome as mRS ≥3
good functional outcome at 3 months | 3 months
  good functional outcomes as mRS≤2; poor outcome as mRS ≥3

CONTACTS AND LOCATIONS:
Overall Officials: zhu Shi, PhD,MD, Principal Investigator — dongguan peoples' hospital
Locations (1):
- Dongguan Peoples' Hospital, Dongguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Under regulations of local ethic committee, data concerning individual privacy are not allowed to release.

REFERENCES:
- [Derived] Shi Z, Li ES, Zhong JS, Yuan JL, Li LR, Zheng CW. Predictive Significance of Day-to-Day Blood Pressure Variability in Acute Ischemic Stroke for 12-Month Functional Outcomes. Am J Hypertens. 2017 May 1;30(5):524-531. doi: 10.1093/ajh/hpx005. PMID 28203689